CLINICAL TRIAL: NCT00091104
Title: A Study in Metastatic Melanoma Using a Lymphodepleting Conditioning Followed by Infusion of Anti-MART-1 TCR-Gene Engineered Lymphocytes and Subsequent Peptide Immunization
Brief Title: Cyclophosphamide and Fludarabine Followed by Vaccine Therapy, Gene-Modified White Blood Cell Infusions, and Aldesleukin in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 040251; 04-C-0251; NCI-6974; CDR0000383246; NCT00088439 (obsolete NCT alias)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Filgrastim; incomplete Freund's adjuvant; Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation

INTERVENTIONS:
Biological: MART-1:27-35 peptide vaccine
Biological: aldesleukin
Biological: filgrastim
Biological: incomplete Freund's adjuvant
Biological: therapeutic autologous lymphocytes
Biological: therapeutic tumor infiltrating lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate
Procedure: autologous hematopoietic stem cell transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Inserting a laboratory-treated gene into a person's white blood cells may make the body build an immune response to kill tumor cells. Giving cyclophosphamide and fludarabine before a white blood cell infusion may suppress the immune system and allow tumor cells to be killed. Vaccines may make the body build an immune response to kill tumor cells. Aldesleukin may stimulate a person's white blood cells to kill tumor cells. Combining white blood cell infusion with vaccine therapy and aldesleukin may cause a stronger immune response and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gene-modified white blood cells when given together with cyclophosphamide, fludarabine, vaccine therapy, and aldesleukin and to see how well it works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of peripheral blood lymphocytes (PBLs) retrovirally transduced with an anti-MART-1 T-cell receptor (TCR) gene followed by high-dose aldesleukin (IL-2) and MART-1:27-35 peptide vaccine in patients with HLA-A*0201-positive metastatic melanoma receiving a myeloablative preparative regimen comprising cyclophosphamide, fludarabine phosphate, and total-body irradiation.
* Determine, preliminarily, whether antitumor antigen TCR-engineered tumor-infiltrating lymphocytes or PBLs followed by IL-2 and MART-1:26-35 after a nonmyeloablative but lymphoid-depleting preparative regimen will result in clinical tumor regression in these patients.

Secondary

* Determine the in vivo survival of TCR gene-engineered cells from these patients.
* Evaluate, preliminarily, clinical response in these patients.

OUTLINE: Patients with resectable tumor undergo tumor biopsy. Tumor-infiltrating lymphocytes (TILs) from the tumor sample are cultured in vitro and tested for reactivity to melanoma antigens. Patients who are unable to undergo biopsy or whose TILs do not grow in culture are assigned to groups I or II. Patients whose tumors yield TILs that do not exhibit melanoma reactivity are assigned to group III. Patients with TILs that exhibit melanoma reactivity are removed from the study.

* Autologous stem cell collection: Patients undergo stem cell collection on treatment protocol NCI-03-C-0277 for reinfusion after the myeloablation and cell therapy. Patients receive filgrastim (G-CSF) subcutaneously (SC) twice daily beginning on day 0 and continuing for up to 5 days. Patients then undergo stem cell collection by apheresis or bone marrow harvest beginning on day 5 and continuing for up to 3 days. Some patients may receive a second course of G-CSF and undergo additional stem cell collection by apheresis or undergo treatment as outlined in group II.
* Group I (peripheral blood lymphocytes [PBLs] with myeloablative preparative regimen): Patients receive a myeloablative preparative regimen comprising cyclophosphamide IV over 1 hour on days -7 and -6, fludarabine phosphate IV over 15-30 minutes on days -7 to -3, and total-body irradiation twice daily on days -3 to -1. Patients also receive autologous in vitro tumor-reactive, T-cell receptor (TCR) gene-transduced PBLs IV over 20-30 minutes on day 1 and aldesleukin IV over 15 minutes every 8 hours on days 1-5, and G-CSF SC daily beginning on day 1 and continuing until blood counts recover.
* Group II (PBLs with nonmyeloablative preparative regimen): Patients who do not meet the eligibility criteria for group I receive a nonmyeloablative preparative regimen comprising cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine phosphate IV over 30 minutes on days -5 to -1. Patients then receive aldesleukin, and G-CSF as in group I.
* Group III (autologous transduced TILs): Patients who have resected tumors that yield viable TILs have their TILs transduced with the anti-MART-1 TCR gene retroviral vector. Patients receive cyclophosphamide and fludarabine phosphate as in group II. Patients then receive autologous transduced TILs IV over 20-30 minutes on day 0. Patients also receive G-CSF and high-dose aldesleukin as in group I.

All patients receive peptide immunizations with MART-1:27-35 peptide vaccine emulsified in incomplete Freund's adjuvant SC on days 0-4, 11, 18, and 25.

In groups II or III, treatment may repeat once 6-8 weeks later for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Treatment may consist of the first type cell infusion or patients may crossover to receive the other cell infusion (PBLs vs TILs).

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 136 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma
* HLA-A*0201-positive disease
* Measurable disease
* Refractory to standard therapy, including high-dose aldesleukin therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* Lymphocyte count > 500/mm^3
* WBC > 3,000/mm^3
* No coagulation disorder

Hepatic

* ALT and AST < 3 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL for patients with Gilbert's disease)
* Hepatitis B antigen negative
* Hepatitis C antibody negative (unless antigen negative)

Renal

* Creatinine ≤ 1.6 mg/dL

Cardiovascular

* No myocardial infarction
* No cardiac arrhythmias
* No cardiac ischemia
* LVEF ≥ 45% by stress cardiac test* (for patients ≥ 50 years of age OR those with a history of EKG abnormalities)
* No other major cardiovascular illness by stress thallium or comparable test NOTE: *Stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test

Pulmonary

* No major respiratory illness
* No obstructive or restrictive pulmonary disease
* FEV_1 ≥ 60% of predicted on pulmonary function test*
* DLCO ≥ 60% predicted (for total-body irradiation cohort) NOTE: *For patients with a prolonged history of cigarette smoking or symptoms of respiratory dysfunction

Immunologic

* HIV negative
* No major immune system illness
* No active systemic infection or opportunistic infection
* No primary immunodeficiency (e.g., autoimmune colitis or Crohn's disease)
* No secondary immunodeficiency (e.g., due to chemotherapy or radiotherapy)
* No history of severe immediate hypersensitivity reaction to study drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after completion of study treatment
* Must sign a durable power of attorney

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* Recovered from prior immunotherapy
* Prior immunization to melanoma antigens allowed

  * Progressive disease during prior immunization allowed
* Prior cellular therapy, including vector transduction with or without myeloablation, allowed
* More than 6 weeks since prior anticytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) monoclonal antibody (MDX-010) therapy
* No prior anti-CTLA-4 antibody unless a post anti-CTLA-4 antibody treatment colonoscopy was normal by biopsy

Chemotherapy

* Recovered from prior chemotherapy

Endocrine therapy

* No concurrent systemic steroids

Radiotherapy

* Recovered from prior radiotherapy
* No prior significant mediastinal or lung radiation (for total-body irradiation cohort)

Surgery

* Not specified

Other

* More than 4 weeks since prior systemic therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2004-07; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety
Tumor regression

SECONDARY OUTCOMES:
In vivo survival of transplanted cells
Clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland